CLINICAL TRIAL: NCT07235748
Title: A Phase 1, Open-label, Single-sequence, 2-period Study to Evaluate the Effect of Multiple Doses of Vorasidenib on the Pharmacokinetics of a Single Dose of Sensitive Index Substrates of Cytochrome P450 2B6, 2C8, 2C9, 2C19, 3A4, and Breast Cancer Resistance Protein in Healthy Adult Participants
Brief Title: Drug-drug Interaction Study of Vorasidenib With Bupropion, Repaglinide, Flurbiprofen, Omeprazole, Midazolam, and Rosuvastatin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S095032-230
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants
MeSH Terms: interventions — vorasidenib; Bupropion; Flurbiprofen; Omeprazole; Midazolam; repaglinide; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vorasidenib and cytochrome P450 and transporter index substrates (Experimental): Participants will receive a single oral dose of 50mg flurbiprofen, 20mg omeprazole, 2mg midazolam and 0.5mg repaglinide on Day 1, 150mg bupropion on Day 2, and 10mg rosuvastatin on Day 5.
  Participants will receive an oral daily dose of 40mg vorasidenib from Day 8 to Day 28. In addition, participants will receive a single oral dose of 50mg flurbiprofen, 20mg omeprazole, 2mg midazolam and 0.5mg repaglinide on Day 22, 150mg bupropion on Day 23, and 10mg rosuvastatin on Day 26, co-administered with vorasidenib.
  Interventions: Drug: Vorasidenib; Drug: Bupropion; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam; Drug: Repaglinide; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Vorasidenib — 40mg taken orally daily from Day 8 through Day 28
Drug: Bupropion — 150mg taken orally on Day 2 and Day 23
Drug: Flurbiprofen — 50mg taken orally on Day 1 and Day 22
Drug: Omeprazole — 20mg taken orally on Day 1 and Day 22
Drug: Midazolam — 2mg taken orally on Day 1 and Day 22
Drug: Repaglinide — 0.5mg taken orally on Day 1 and Day 22
Drug: Rosuvastatin — 10mg taken orally on Day 5 and Day 26

SUMMARY:
The objective of this study is to evaluate the effect of multiple doses of vorasidenib on single-dose PK of bupropion as an index substrate of CYP2B6, flurbiprofen as an index substrate of CYP2C9, omeprazole as an index substrate of CYP2C19, repaglinide as an index substrate of CYP2C8, midazolam as an index substrate of CYP3A4, and rosuvastatin as a substrate of BCRP in healthy adult participants. The study consists of screening, two treatment periods in-house, and a follow-up period. During the first period, Day 1 through Day 7, participants will receive CYPs and BCRP index substrates alone and during the second treatment period, Day 8 through Day 28, these will be administered in combination with vorasidenib. Participation in the study will be up to 87 days from screening through the follow up period.

Study activities may include blood tests, ECG, vital signs, and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-lactating female participants, including women of childbearing potential (WOCBP).
* Body mass index (BMI) of 18.0 - 30.0 kg/m² (both inclusive), at Screening.
* Body weight of at least 40 kg, at Screening.
* Female participants of childbearing potential must use 2 effective methods of birth control, or abstinence from Screening until at least 90 days after the last dose of vorasidenib; be surgically sterile at least 6 months prior to the first dose of investigational medicinal product (IMP) in the study; or be postmenopausal. Female participants of childbearing potential must have a negative serum pregnancy test at Screening and prior to the first dose of IMP in the study.
* Male participants with female partners of childbearing potential must be sterile, be willing to use 2 effective methods of birth control from Screening until at least 90 days after the last dose of vorasidenib, or practice abstinence from Screening until at least 90 days after the last dose of vorasidenib. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the participant. Male participants should also agree to not donate sperm for the duration of the study and until at least 90 days after the last dose of vorasidenib.
* The participant is a continuous nonsmoker who has not used nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) for at least 3 months prior to the first dose of IMP in the study based on a cotinine test result.
* The participant is considered by the investigator (or designee, if applicable) to be in good general health as determined by medical history, full physical examination, clinical laboratory test results, 12-lead electrocardiogram (ECG) results, and vital sign measurements findings at screening and admission.

Exclusion Criteria:

* The participant is a WOCBP who is pregnant, lactating, or planning to become pregnant within at least 90 days after the last dose of vorasidenib in the study; the participant is on oral contraceptive pills or contraceptive patch within 14 days or 5 half-lives (whichever is longer) prior to the first dose of IMP in the study; the participant used a hormonal IUD or vaginal ring within 3 months prior to the first dose of IMP in the study; or the participant received any injectable or implantable hormone-containing product within 1 year prior to the first dose of IMP in the study.
* The participant has consumed grapefruit or grapefruit juice or Seville orange or Seville orange-containing products (e.g., marmalade) within 14 days prior to the first dose of IMP in the study.
* The participant has ingested vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard) and charbroiled meats within 14 days prior to the first dose of IMP in the study.
* The participant has consumed caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate), alcohol, or products containing any of these within 48 hours prior to the first dose of IMP in the study.
* The participant is unable or unwilling to abstain from recreational drugs, alcohol, caffeine, xanthine-containing beverages or food (e.g., coffee, tea, chocolate, and caffeinated sodas, colas), grapefruit, grapefruit juice, Seville oranges, or products containing any of these, from 48 hours (caffeine, xanthine-containing beverages or food, alcohol) or 14 days (recreational drugs, grapefruit, grapefruit juice, Seville oranges, or Seville orange-containing products) prior to the first dose of IMP in the study until the Discharge/Early Termination visit.
* The participant has received any vaccine or used any prescription (including hormonal birth control or hormone replacement therapy) or over-the-counter medications (except acetaminophen/paracetamol [up to 2 g per 24 hours] or ibuprofen [up to 1.2 g per 24 hours]), including herbal (e.g., St. John's Wort) or nutritional supplements, within 14 days or 5 drug half-lives, whichever is longer, prior to the first dose of IMP in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration (AUC0-last) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Area under the plasma concentration versus time curve from 0 extrapolated to infinity (AUC0-inf) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Time corresponding to Cmax (Tmax) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Terminal half-life (t1/2) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Apparent oral clearance (CL/F) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Apparent volume of distribution during the terminal phase following oral administration (Vz/F) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29
Elimination rate constant (Kel) of bupropion and its metabolite hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, and rosuvastatin | Through Day 29

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | Through the Follow-up Phone Call (Day 57)
Trough plasma concentration (Ctrough) of vorasidenib | Through Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/